CLINICAL TRIAL: NCT03021109
Title: Assessment of Volume Status by Measurement of Caval Index by Bedside Ultrasound in Children With Acute Gastroenteritis
Brief Title: Assessment of Volume Status by Bedside Ultrasound in Children With Acute Gastroenteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ASIM ENES ÖZBEK, Emergency medicine specialist, Derince Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/278
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Dehydration; Acute Gastroenteritis
Keywords: ultrasound; pediatrics; gastroenteritis
MeSH Terms: conditions — Dehydration; Gastroenteritis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inferior vena cava diameteres (Experimental): Measurement of inferior vena cava diameters with ultrasound
  Interventions: Device: Measurement of inferior vena cava diameters with ultrasound

INTERVENTIONS:
Device: Measurement of inferior vena cava diameters with ultrasound — The patient is placed in the supine position. Curvilinear probe is used. Subxiphoid view is obtained. The IVC is visualized in the longitudinal plane as it enters the right atrium. The diameter of the IVC for calculation of the caval index is measured 2 cm from where it enters the right atrium

SUMMARY:
The purpose of the study is assessment of volume status by bedside ultrasound in children with acute gastroenteritis

DETAILED DESCRIPTION:
The research will be conducted of emergency medicine department in the Derince Training and Research Hospital. Patients referred to acute gastroenteritis will be included to the study. After initial evaluation, the clinician will inform the principal investigator about the patient. The principal investigator will record the patient's demographic data, contact information, vital signs, history, physical examination findings, and weight. Than expirium and inspirium diameters of vena cava inferior will be measured with the bedside ultrasound and caval index will be calculated. An investigator who have had an ultrasound certification by Emergency Medicine Association of Turkey for six years will make the measurements. After 1 week the patient will called up for re-evaluation. Applicants' weights will be measured again with the same weighing machine. The differences between initial and after one week weight measurement will be accepted as the gold standard method for volume loss. The weight loss of the patient, the dehydration findings detected on physical examination and the caval index will be compared.

Data will be collected on predesigned data sheets, by an investigator and subsequently will be entered into a spreadsheet (Excel 2007; Microsoft, Redmond, WA). All recorded data will be checked by an another investigator to identify possible errors. Results will be submitted at least every two months.

Linear regression will be performed with dehydration as the dependent variable and the caval index as the independent variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 6 months and 18 years of age who presented to the Emergency Department with gastroenteritis

Exclusion Criteria:

* congenital heart disease
* chronic liver disease
* chronic renal disease
* patients or parents who doesn't want to enroll the study

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
The correlation of caval index with the amount of fluid loss in pediatric patients with acute gastroenteritis | 1 week

SECONDARY OUTCOMES:
The correlation between physical examination findings and the amount of fluid loss in pediatric dehydration | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Asım E. Özbek, Specialist, Principal Investigator — Kocaeli Derince Training and Research Hospital
Locations (1):
- Kocaeli Derince Training and Research Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van den Berg J, Berger MY. Guidelines on acute gastroenteritis in children: a critical appraisal of their quality and applicability in primary care. BMC Fam Pract. 2011 Dec 2;12:134. doi: 10.1186/1471-2296-12-134. PMID 22136388
- [Background] Liebelt EL. Clinical and laboratory evaluation and management of children with vomiting, diarrhea, and dehydration. Curr Opin Pediatr. 1998 Oct;10(5):461-9. doi: 10.1097/00008480-199810000-00002. PMID 9818241
- [Background] Steiner MJ, DeWalt DA, Byerley JS. Is this child dehydrated? JAMA. 2004 Jun 9;291(22):2746-54. doi: 10.1001/jama.291.22.2746. PMID 15187057
- [Background] McConnochie KM, Conners GP, Lu E, Wilson C. How commonly are children hospitalized for dehydration eligible for care in alternative settings? Arch Pediatr Adolesc Med. 1999 Dec;153(12):1233-41. doi: 10.1001/archpedi.153.12.1233. PMID 10591299
- [Background] Haciomeroglu P, Ozkaya O, Gunal N, Baysal K. Venous collapsibility index changes in children on dialysis. Nephrology (Carlton). 2007 Apr;12(2):135-9. doi: 10.1111/j.1440-1797.2006.00700.x. PMID 17371335
- See also: Related Info — http://www.who.int/mediacentre/factsheets/fs330/en/